CLINICAL TRIAL: NCT03497455
Title: Feasibility Study to Evaluate Utility of the BARCO NV Digital Dermatoscope in the Skin Cancer Clinic
Brief Title: Utility of Digital Dermoscopy in the Skin Cancer Clinic
Status: Terminated | Type: Observational
Why Stopped: COVID pandemic / Change in strategic direction
Sponsor: Barco NV (Industry)
Responsible Party: Sponsor
Other Study IDs: 234237
Record Dates: First submitted 2018-04-05; First posted 2018-04-13 (Actual); Last update posted 2021-12-29 (Actual); Status verified 2021-12

CONDITIONS: Skin Cancer; Dermatology/Skin - Other
MeSH Terms: conditions — Skin Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Barco NV Digital Dermatoscope device images — Images taken by Clinician in consultation OR in Dermatology department theatres OR images taken in medical photography suite - in the latter case, images can be taken by medical photographer or Research nurse or Dermatologist
Device: Standard medical photographs including dermoscopy images — Images taken by medical photographer as part of standard care in the medical photography suite.
Other: Clinic proforma completion — This is part of standard care and will be undertaken by the clinician who is responsible for the patient

SUMMARY:
This feasibility study aims to evaluate the use of the BARCO NV digital dermatoscope (non-CE marked device) in the skin cancer clinic. All eligible patients attending the Dermatology outpatient skin cancer clinic will be invited to participate. Patients who consent to the study will undergo standard care which will include medical photography of skin lesion(s) and appropriate management as determined by the Consultant Dermatologist in clinic. In addition to standard care, patients will undergo photography of the same lesion(s) using the BARCO NV digital dermatoscope. There will be no other intervention and no additional hospital visits in relation to the study. Use of the device will not influence the clinical management of the patient.

A detailed experience questionnaire will be administered to all clinicians using the BARCO device to explore their opinion on its ease of use and features.

All standard macroscopic & dermoscopic images will be taken by OUH medical illustration department and stored on the 'Fotoweb' database (in keeping with current standard practice). Trained Dermatology Consultants, Dermatology Registrars, Research nurses or Medical Photographers, will take BARCO NV device images. A database of all BARCO images will be collected and stored on a dedicated NHS computer separate from the patient clinical record. Standard medical photography images will be stored on Fotoweb as per standard NHS clinical care.

Data will be anonymised and collated and then sent securely to BARCO for further analyses to enable optimization of the BARCO device and for development of diagnostic algorithms in the future.

ELIGIBILITY:
Inclusion Criteria:

* Participant is willing and able to give informed consent for participation in the study.
* Male or Female, aged 18 years or above.
* Patient presenting with any visible skin lesion for Dermatologist review on a body site amenable for optimal photographic imaging
* Able and willing to comply with all study requirements.
* Patient with a skin lesion that is clinically diagnosed by a Consultant Dermatologist as benign OR a suspicious skin lesion requiring excisional biopsy for histological diagnosis
* Patient attending for a 'New' or 'Follow-up' consultation

Exclusion Criteria:

* Patients aged under 18 years old
* Patients unable to provide informed consent
* Skin lesions in an anatomical site which is not suitable for photography including genital lesion, hair-bearing site or subungual lesion
* Maximum size of lesion 25 mm
* Lesion is at a site where previous surgery was undertaken
* Lesion on a mucosal site

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: All eligible & consenting participants will be approached in a Skin Cancer clinic. Once the clinic consultation has been completed and a decision regarding their management has been made, patients will be invited to consent to the study.
Sampling Method: Non-Probability Sample
Enrollment: 13 (Actual)
Dates: Start 2018-07-12 (Actual); Primary Completion 2020-03-17 (Actual); Study Completion 2020-03-17 (Actual)

PRIMARY OUTCOMES:
Clinician experience questionnaire results | 1 year
  To assess the acceptability of the new dermoscope in the skin cancer clinic, questions about the usability of the device and about the image quality of the obtained dermoscopic pictures are included.

SECONDARY OUTCOMES:
Collection of image database | 1 year
  Anonymised database of clinicopathological and digital images of benign, malignant and equivocal skin lesions + Proportion of high quality images amenable to clinician evaluation
Safety of the device for the patient and the user: occurrence of adverse events | 1 year
  Number of adverse events reported

CONTACTS AND LOCATIONS:
Locations (1):
- Oxford University Hospitals NHS Foundation Trust, Oxford, United Kingdom